CLINICAL TRIAL: NCT07279051
Title: Modified Mini-Open TLIF Versus Traditional Open TLIF for Lumbar Spinal Stenosis : A Prospective, Randomized Controlled Trial
Brief Title: Modified Mini-Open TLIF vs Traditional Open TLIF
Acronym: TLIF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY-20250801001-02
Record Dates: First submitted 2025-11-16; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Spinal Stenosis Lumbar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mMO-TLIF surgery group (Experimental): The experimental group (mMO-TLIF group) underwent modified Mini-Open Transforminal Lumbar Interbody Fusion, a procedure performed under general anesthesia via a posterior minimally invasive approach through the transforminal corridor. Key steps involved dilating the paraspinal musculature unilaterally with a retractor following exposure, subsequently performing pedicle screw insertion, decompression, and interbody cage placement, supplemented by contralateral percutaneous pedicle screw fixation.
  Interventions: Procedure: modified mini-open transforaminal lumbar interbody fusion
- Traditional TLIF surgery group (Active Comparator): The traditional Open Transforminal Lumbar Interbody Fusion (TLIF) is a classic spinal surgical procedure. It is characterized by a long midline open incision, which requires extensive subperiosteal dissection and stripping of the paraspinal muscles to expose the bony anatomy. This approach provides a wide, direct surgical field, allowing for pedicle screw placement, neural decompression, and interbody fusion to be performed under direct visualization.
  Interventions: Procedure: traditional transforaminal lumbar interbody fusion

INTERVENTIONS:
Procedure: modified mini-open transforaminal lumbar interbody fusion — The modified Mini-Open Transforaminal Lumbar Interbody Fusion (mMO-TLIF) is a hybrid technique that integrates minimally invasive and open concepts. Its core principle involves a limited open exposure on the decompression side for canal decompression and interbody fusion using retractors, while the non-decompression side undergoes pure percutaneous pedicle screw fixation, thereby maximally preserving the paraspinal muscles. This approach effectively balances surgical visualization with tissue preservation, achieving robust internal fixation while significantly reducing muscle injury, intraoperative blood loss, and enhancing surgical efficiency, making it particularly suitable for multi-level fusion.
  Arms: mMO-TLIF surgery group
Procedure: traditional transforaminal lumbar interbody fusion — Traditional Transforaminal Lumbar Interbody Fusion (TLIF) is a classic posterior surgical approach for lumbar pathologies. It utilizes a posterior midline incision with extensive dissection and retraction of paraspinal muscles to achieve adequate exposure, allowing for discectomy, neural decompression, and interbody fusion through a unilateral transforaminal approach, typically supplemented with bilateral pedicle screw instrumentation.
  Advantages: Excellent surgical exposure and large working space facilitating thorough neural decompression and providing reliable spinal stability.
  Disadvantages: Extensive dissection of paraspinal soft tissues may lead to postoperative chronic muscle denervation and low back pain; associated with significant intraoperative blood loss and a prolonged recovery period.
  Arms: Traditional TLIF surgery group

SUMMARY:
This clinical study aims to find out if a modified mini-open spine surgery (modified mini-open transforaminal lumbar interbody fusion，mMO-TLIF) is as good as, or better than, the traditional open surgery (traditional transforaminal lumbar interbody fusion，traditional TLIF) for treating low back pain, leg pain, and walking difficulties caused by lumbar spinal stenosis with instability. The study will also look at the safety of both surgeries.

It is designed to answer these main questions:

Is the mMO-TLIF surgery as good as the traditional TLIF surgery at improving patients' lower back function and quality of life? Does the mMO-TLIF surgery reduce blood loss during the operation and shorten hospital stays and recovery time? What medical problems (like infections or nerve injuries) might patients experience after having the mMO-TLIF surgery? Researchers will compare the results of the mMO-TLIF surgery group with the traditional TLIF surgery group to see which one works better.

Participants will:

Be randomly assigned to receive either the mMO-TLIF minimally invasive surgery or the traditional TLIF open surgery.

Come back to the hospital for check-ups before surgery, and then at 1 month, 3 months, 12 months and 24 months after surgery.

During these check-ups, they will have physical exams, fill out questionnaires about their symptoms, dysfunction and quality of life, and get X-rays or CT scans to see how their bones are healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years.
* Presence of unilateral neurogenic claudication or radicular pain in the lower limbs, with failure to respond to at least 3 months of conservative treatment.
* Presence of bilateral neurogenic claudication or radicular pain in the lower limbs, but with complete resolution of neurological symptoms in at least one lower limb during recumbency and an unremarkable physical examination, alongside failure to respond to at least 3 months of conservative treatment.
* Radiologically confirmed single- or two-level lumbar spinal stenosis on MRI, with evidence of instability specifically at the stenotic level(s) on standing lateral radiographs.
* The mMO-TLIF or TLIF surgical procedure is performed by the same lead surgeon at each participating investigational site.
* Subjects voluntarily participate and provide written informed consent.

Exclusion Criteria:

* Presence of bilateral radicular pain in the lower limbs that does not completely resolve at rest.
* History of previous lumbar spine trauma or surgery.
* Presence of spinal infection, tuberculosis, or tumor.
* Contraindications to surgery, such as severe systemic medical diseases, coagulation disorders, severe active infectious diseases, or osteoporosis.
* Significant intervertebral space collapse, presence of bony ankylosis, etc.
* Incomplete data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-12-06 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | preoperatively and 1/3/12/24 months postoperatively
  Oswestry Disability Index (ODI), a 10-item questionnaire scored from 0 (no disability) to 100 (maximum disability), with higher scores indicating worse disability.

SECONDARY OUTCOMES:
Pain VAS scores | preoperatively and 1/3/12/24 months postoperatively
  Pain Visual Analog Scale (VAS) score, ranging from 0 (no pain) to 10 (worst pain), with higher scores indicating more severe pain.
Zurich Claudication Questionnaire (ZCQ) score | Preoperative and 1/3/12 months postoperative
  Zurich Claudication Questionnaire (ZCQ) score, which includes symptom severity (range 1 to 5, lower scores indicate milder symptoms) and physical function (range 1 to 5, lower scores indicate less disability).
Brock Quality of Life Five Dimensions (EQ-5D-3L) questionnaire score | 1/24 month postoperatively
  EuroQol 5-Dimension 3-Level (EQ-5D-3L) questionnaire score, ranging from -0.59 to 1.0, with higher scores indicating better quality of life.
Operative Time | Immediately upon surgery conclusion
  Operative Time, measured in minutes
Intraoperative Blood Loss | Immediately upon surgery conclusion
  Intraoperative Blood Loss, measured in milliliters
Transfusion Rate | From surgery start until hospital discharge, assessed up to 30 days.
Time to Ambulation | Time from surgery to first ambulation, assessed during postoperative hospital stay up to 30 days
Length of Hospital Stay | Length of hospital stay from surgery to discharge, assessed up to 30 days.
Incidence of complications | From surgery start until 24 months postoperatively.
  e.g., nerve injury, infection, screw loosening
Radiographic fusion rate | 12 months postoperative
  Evaluated by CT (Bridwell classification)

IPD SHARING:
Plan to Share IPD: No